CLINICAL TRIAL: NCT06034730
Title: Breathomics: May it Become an Affordable, New Tool for Early Diagnosis and Screening of Lung Cancer? An Exploratory Study on a Cohort of 60 Patients
Brief Title: Breathomics: May it Become an Affordable, New Tool for Early Diagnosis and Screening of Lung Cancer?
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: University of Michigan (Other); Humanitas Hospital, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: 665139
Record Dates: First submitted 2023-09-01; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer
Keywords: breathomic; NSCLC; screening; volatile organic compounds
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breath from the patients, retained for a maximum of 24h
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung Cancer Patients: patients undergoing surgery for histologically proven NSCLC
  Interventions: Device: Portable GC device for brath analysis
- Healthy Control Patients: patients undergoing surgery for benign extra-thoracic disease who had undergone chest X-rays/chest CT-scan, proved to be negative during preoperative evaluation.
  Interventions: Device: Portable GC device for brath analysis

INTERVENTIONS:
Device: Portable GC device for brath analysis — Patients were asked to orally exhale 1-2 L breath into a 5 L Tedlar bag via a one-way mouthpiece and Nafion filter for moisture removal, as shown in Figure 1B. The process usually takes about a few minutes. The breath analysis took place either in-situ immediately after the breath sample collection or within 24 h of breath collection. The Tedlar bags were stored under ambient condition until analyzed. During the breath analysis, the Tedlar bag was connected to the sampling port of the portable GC (Figure 1C). Approximately 350 mL of breath was pulled from the Tedlar bag into the GC for analysis. The GC operation was controlled using LabView via a laptop. The total assay time was 30 min, including 5 min of breath sampling time from the Tedlar bag at a flow rate of 70 mL/min (see the blue path in Figure 1A), 5 min of desorption/transfer time, 10 min of chromatographic separation time (see the orange path in Figure 1A), and 10 min of GC system cleaning time.

SUMMARY:
Breath analysis examining specific patterns of volatile organic compounds (VOCs) has been demonstrated to be able to discriminate lung cancer (LC) patients from healthy controls (HC). However, the existing technology uses complex, expensive, and low throughput analytical platforms to give an offline response, thus preventing its applicability for mass screening. The reliability of a new portable device to enable rapid, on-site LC diagnosis is tested.

DETAILED DESCRIPTION:
The breath of patients with histologically proven NSCLC and healthy controls was sampled into Tedlar bags through a Nafion filter and a one-way mouthpiece. The breath samples in the bags were then analyzed by an automated micro portable gas chromatography device developed in-house, which consisted of a thermal desorption tube, thermal injector, separation column, and photoionization detector, as well as other accessories such as pumps, valves, and a helium cartridge. The chromatograms were analyzed by chemometrics and machine learning techniques.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC histologically proven (for LC group) at any stage of disease
* non-cancer controls who had negative findings on preoperative chest X-rays/chest CT scan (for HC groups)

Exclusion Criteria:

* Patients who had any history of another type of cancer
* who had received neoadjuvant chemo/radiotherapy because of the possible unknown effects on cancer metabolism
* pediatric patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 60 patients undergoing surgery for histologically proven NSCLC and a comparative group of non-cancer controls who had negative findings on preoperative chest X-rays/chest CT scan were admitted to our Thoracic Surgery Unit between August 2021 and March 2022. Patients underwent breath collection during the pre-hospitalization analysis before surgery. The control group was recruited from patients undergoing surgery for benign extra-thoracic disease who had undergone chest X-rays/chest CT-scan, proved to be negative during preoperative evaluation.
  Patients excluded from analysis were those who had any history of another type of cancer and those who had received neoadjuvant chemo/radiotherapy because of the possible unknown effects on cancer metabolism.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Changes in VOCs peaks in patients with lung cancer vs healthy patients | 24 hours
  Identify biomarkers able to discriminate between lung cancer patients and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Marulli, MD, PhD, Study Director — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- Azienda Consorziale Ospedaliero-Universitaria Policlinico di Bari - Thoracic Surgery Unit, Bari, Italy

IPD SHARING:
Plan to Share IPD: No
On request alla data will be available

REFERENCES:
- [Derived] Brascia D, De Iaco G, Panza T, Signore F, Carleo G, Zang W, Sharma R, Riahi P, Scott J, Fan X, Marulli G. Breathomics: may it become an affordable, new tool for early diagnosis of non-small-cell lung cancer? An exploratory study on a cohort of 60 patients. Interdiscip Cardiovasc Thorac Surg. 2024 Sep 4;39(3):ivae149. doi: 10.1093/icvts/ivae149. PMID 39226187